CLINICAL TRIAL: NCT06136767
Title: Registry for Systemic Eczema Treatments
Acronym: RESET
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Doris Duke Charitable Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00372852
Record Dates: First submitted 2023-11-06; First posted 2023-11-18 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 26 Years
Biospecimen Retention: Samples With DNA — Biospecimen collection is voluntary and may include:
  1. Skin Biopsies: a small punch biopsy (3-4mm) or shave biopsy (around 1 cm).
  2. Blood Samples: 2-5 teaspoons may be collected depending on the participant's weight.
  3. Skin Swabs: Skin swabs may be collected from a target area of the skin to study the microbiome.
  4. Buccal (cheek) Swabs: Buccal swabs may be collected from the inner cheek to collect cheek cells.
  5. Tape Stripping: Tape strips may be collected from a target area of the skin.
  6. Hair Samples: Hair may be collected from up to 5 various regions.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Methotrexate: Participants who have received methotrexate for atopic dermatitis.
- Cyclosporine: Participants who have received cyclosporine for atopic dermatitis.
- Mycophenolate mofetil: Participants who have received mycophenolate mofetil for atopic dermatitis.
- Azathioprine: Participants who have received azathioprine for atopic dermatitis.
- Dupilumab: Participants who have received dupilumab for atopic dermatitis.
- Tralokinumab: Participants who have received tralokinumab for atopic dermatitis.
- Upadacitinib: Participants who have received upadacitinib for atopic dermatitis.
- Abrocitinib: Participants who have received abrocitinib for atopic dermatitis.

SUMMARY:
The Registry for Systemic Eczema Therapies (RESET) registry is a database and biospecimen repository for patients with pediatric-onset atopic dermatitis (AD) who have used or will initiate any systemic treatment(s) for AD. The goal of the registry is to enable more efficient research recruitment and data collection as well as timely notification to enrollees about newly FDA-approved treatments for AD.

DETAILED DESCRIPTION:
The purpose of the Registry for Systemic Eczema Therapies (RESET) registry is to serve as a database and biospecimen repository of patients with pediatric-onset atopic dermatitis (AD), also known as eczema. This registry seeks to enroll patients with AD who have used or will initiate any systemic treatment(s) for AD. Such a registry will allow investigators to identify patients who are potentially eligible for AD research protocols, including observational studies or clinical trials. The registry will also prospectively collect data that would then serve as a resource for studying a variety of questions surrounding systemic therapy use in patients with AD, for example comparing the effectiveness of treatments or examining treatment effects on patient-reported outcomes. Moreover, the registry would permit safety monitoring of systemic AD medications, as it would include both patients receiving traditional systemic agents with well-known side effect profiles and patients receiving more novel systemic agents with under-characterized side effect profiles. Finally, this registry would allow for the identification of patients with moderate-to-severe AD who may be eligible to receive and benefit from the rapidly expanding number of U.S. Food and Drug Administration (FDA)-approved systemic therapies for AD.

ELIGIBILITY:
Inclusion criteria:

* Age <26 years old
* Current physician diagnosis of atopic dermatitis
* Provide signed informed consent if ≥ 18 years old
* Provide signed informed consent by parent or legal guardian (if <18 years old) and informed assent if applicable
* Subject and/or parent/legal guardian is willing to be contacted in the future by study staff
* Seen for clinical care at Johns Hopkins since 1/1/2017
* Previously on, currently on, or planning to initiate (within next 6 months) a systemic AD therapy

Exclusion criteria:

* Age ≥26 years old at the time of registry enrollment
* Does not speak English
* If <18 years old, has a primary caretaker who does not speak English
* If <18 years old, parent/legal guardian is unwilling to sign the written informed consent
* Is a foster child
* Has not received clinical care at Johns Hopkins since 1/1/2017

Ages: 1 Year to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients with atopic dermatitis treated with systemic therapy for AD and meet the inclusion criteria will be asked to participate in this registry
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-01-17 (Actual); Primary Completion 2030-08-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment effectiveness as assessed by the change in Investigator's Global Assessment (IGA) Scores | 3 years
  To evaluate the clinical effectiveness of systemic treatments for atopic dermatitis according to IGA through periodic electronic medical record (EMR) review. The IGA is a physician-reported atopic dermatitis severity score. IGA is the global clinical assessment scale to determine severity of AD and clinical response to treatment on a static 5-point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on the degree of erythema and papulation/infiltration. The IGA score ranges from 0 to 4. Higher scores indicate greater severity of AD.
Treatment effectiveness as assessed by the change in Eczema Area and Severity Index (EASI) Scores | 3 years
  To evaluate the clinical effectiveness of systemic treatments for atopic dermatitis according to EASI through periodic electronic medical record (EMR) review. The EASI score is a physician-reported atopic dermatitis severity score. EASI is used to evaluate severity of AD based on AD clinical signs and % of body surface area (BSA) affected. Severity of clinical signs of AD (erythema, induration/papulation, excoriation and lichenification) is scored separately for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin] and lower limbs [including buttocks]) on 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. The total EASI score ranges from 0 to 72. Higher scores indicate greater severity of AD.
Treatment effectiveness as assessed by the change in Patient Oriented Eczema Measure (POEM) Scores | Quarterly from baseline to 3 years
  To evaluate the effectiveness of systemic treatments for atopic dermatitis (AD) according to a POEM score. The POEM score is a patient-reported AD severity score. The POEM is a 7-item questionnaire to assess disease symptoms in children and adults with AD. It is composed of 7 items (dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping) based on symptom frequency during the past week (0 = 'no days', 1 = '1 to 2 days', 2 = '3 to 4 days', 3 = '5 to 6' days, and 4 = 'every day'). The total POEM score ranges from 0 to 28. Higher scores indicate more severe disease and poor quality of life.
Treatment effectiveness as assessed by the change in Patient-Reported Outcomes Measurement Information System (PROMIS) Itch questionnaire score | Quarterly from baseline to 3 years
  To evaluate the effectiveness of systemic treatments for atopic dermatitis (AD) according to the PROMIS Itch questionnaire. The PROMIS Itch questionnaire measures the extent to which patients experience problems with itchiness over the past 7 days using a 5-point Likert scale (1 = Never; 2 = Rarely; 3 = Sometimes; 4 = Often; and 5 = Almost Always). Higher scores reflect greater severity of experienced itch symptoms.
Treatment effectiveness as assessed by the change in Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety questionnaire score | Quarterly from baseline to 3 years
  To evaluate the effectiveness of systemic treatments for atopic dermatitis (AD) according to the PROMIS Anxiety questionnaire. The PROMIS Anxiety questionnaire measures the extent to which patients experience problems with anxiety over the past 7 days using a 5-point Likert scale (1 = Never; 2 = Almost never; 3 = Sometimes; 4 = Often; and 5 = Almost Always). The questionnaire includes fear (fearfulness, panic), anxious misery (worry, dread), hyperarousal (tension, nervousness, restlessness), social/separation anxiety (fear or distress when separating from caregivers), and somatic symptoms related to arousal (racing heart, dizziness). Higher scores reflect greater severity of experienced anxiety symptoms.
Treatment effectiveness as assessed by the change in Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Problem questionnaire score | Quarterly from baseline to 3 years
  To evaluate the effectiveness of systemic treatments for atopic dermatitis (AD) according to the PROMIS Sleep Problem/Health questionnaires. The PROMIS Sleep Problem questionnaire measures the extent to which patients experience problems with sleep over the past 7 days using a 5-point Likert scale (1 = Never; 2 = Almost never; 3 = Sometimes; 4 = Almost always; and 5 = Always). The sleep problems contain sleep disturbances (sleep quality, sleep onset, sleep continuity) and sleep-related impairment (perceptions of sleepiness during usual awake hours and reported impairments during the day associated with sleep problems or daytime sleepiness). Higher scores reflect greater severity of sleep problems.
Treatment effectiveness as assessed by the change in Patient-Reported Outcomes Measurement Information System (PROMIS) Depressive Symptoms questionnaire score | Quarterly from baseline to 3 years
  To evaluate the effectiveness of systemic treatments for atopic dermatitis (AD) according to the PROMIS Depressive Symptoms questionnaire. The PROMIS Depressive Symptoms questionnaire measures the extent to which patients experience problems with depression over the past 7 days using a 5-point Likert scale (1 = Never; 2 = Almost never; 3 = Sometimes; 4 = Almost Always; and 5 = Always). The depressive symptoms include negative mood (sadness, guilt), views of self (self-criticism, worthlessness), and social cognition (loneliness, interpersonal alienation); decreased positive affect, anhedonia (loss of interest, inability to engage in play), and engagement. Higher scores reflect greater severity of experienced depressive symptoms.
Treatment effectiveness as assessed by the change in Patient-Reported Outcomes Measurement Information System (PROMIS) Cognitive Function questionnaire score | Quarterly from baseline to 3 years
  To evaluate the effectiveness of systemic treatments for atopic dermatitis (AD) according to the PROMIS Cognitive Function questionnaire. The PROMIS Cognitive Function questionnaire measures the extent to which patients experience problems with cognitive function over the past 4 weeks using a 5-point Likert scale (1 = All of the time; 2 = Most of the time; 3 = Some of the time; 4 = A little of the time; and 5 = None of the time). The questionnaire includes difficulties in cognitive abilities (e.g., memory, attention, and decision making), and difficulties in the application of such abilities to everyday tasks (e.g., planning, organizing, calculating, remembering, and learning). Lower scores reflect greater impact on cognitive function.
Treatment effectiveness as assessed by the change in Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health questionnaire score | Quarterly from baseline to 3 years
  To evaluate the effectiveness of systemic treatments for atopic dermatitis (AD) according to the PROMIS Global Health questionnaire. The PROMIS Global Health questionnaire measures the extent to which patients experience problems with global health in general using a 5-point Likert scale (1 = Poor; 2 = Fair; 3 = Good; 4 = Fair; and 5 = Excellent). The questionnaire includes an overall evaluation of physical, mental health, and social health. Higher scores reflect a lower quality of global health.
Treatment effectiveness as assessed by the change in Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity questionnaire score | Quarterly from baseline to 3 years
  To evaluate the effectiveness of systemic treatments for atopic dermatitis (AD) according to the PROMIS Pain Intensity questionnaire. The PROMIS Pain Intensity questionnaire measures the intensity of patients' pain due to their AD over the past 7 days using a 10 point scale, with 0 indicating "No Pain" and 10 indicating "the worst pain possible." Higher raw scores reflect greater severity of experienced pain due to AD.

SECONDARY OUTCOMES:
Rate of discontinuation or dose de-escalation of systemic treatment | 3 years
  To assess rates of discontinuation or dose de-escalation per systemic treatment (e.g. dupilumab, tralokinumab, upadacitinib and abrocitinib) in patients with well-controlled atopic dermatitis
Adverse effects of systemic treatments for atopic dermatitis | 3 years
  To collect data on adverse effects of systemic treatments for AD (e.g. conjunctivitis, injection site reaction, renal or liver impairment, cardiovascular events, malignancy, infection, etc.) to assess the safety of each systemic treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Joy Wan, MD MSCE, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Background] Laughter MR, Maymone MBC, Mashayekhi S, Arents BWM, Karimkhani C, Langan SM, Dellavalle RP, Flohr C. The global burden of atopic dermatitis: lessons from the Global Burden of Disease Study 1990-2017. Br J Dermatol. 2021 Feb;184(2):304-309. doi: 10.1111/bjd.19580. Epub 2020 Nov 29. PMID 33006135